CLINICAL TRIAL: NCT02068404
Title: Nifedipine Pharmacokinetics and Pharmacodynamics When Used as a Tocolytic in Patients Hospitalized for Acute Threatened Preterm Labour
Brief Title: Nifedipine Pharmacokinetics and Pharmacodynamics When Used as a Tocolytic in Acute Threatened Preterm Labour
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chantal Csajka (Other)
Responsible Party: Sponsor-Investigator, Chantal Csajka, Prof PhD, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK/PD_Nifedipine
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Preterm Labor
Keywords: Tocolysis; Preterm labor; Nifedipine; Pharmacokinetics
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nifedipine (Other)
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Nifedipine
  Other Names: Adalat

SUMMARY:
Preterm birth is the leading cause of perinatal mortality and morbidity. According to WHO, 15 million children are born prematurely (gestational age < 37 weeks) in the world each year while 7% of them die because of complications associated with prematurity. Despite constant improvement of obstetrical care, the number of preterm births has increased over the last decades and prematurity is still the most frequent cause of prenatal hospitalization in industrialized countries.

The American College of Obstetricians and Gynecologists as well as the Royal College of Obstetricians and Gynaecologists recommend nifedipine as a first-line tocolytic in case of acute threatened preterm labour. Clinical experience show however an important variability in treatment response among pregnant women. In spite of its large use in obstetrics as a tocolytic agent, nifedipine is prescribed off-label. As a consequence no international consensus on optimal dose schedule has so far been proposed.

Small sample size and heterogeneousness of tocolysis administration protocols make it difficult to compare the little data available on the pharmacokinetics of nifedipine in pregnant women. Nevertheless an important interindividual variability in concentrations has been identified (CV=12-76%) but very few studies have investigated the possible reasons of this variability in pregnant women. Genetic and environmental factors involved in drug distribution and metabolism (e.g. enzymatic activity, CYP 3A5 genotype) might partially explain variability in drug levels and therefore differences in treatment response.

The goal of this study is to quantify the variability in nifedipine pharmacokinetics and identify potential genetic and non-genetic sources of variability in nifedipine pharmacokinetics in pregnant women. The relationship between concentration and treatment response will be evaluated and will serve to propose optimal dosage regimen to improve efficacy and reduce side effects associated with this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women under nifedipine treatment for acute threatened preterm labour
* Hospitalization for this condition in the maternity of the University Hospital of Lausanne (CHUV)
* Gestational age of 20-34 weeks
* Signed informed consent

Exclusion Criteria:

* Patient < 18 years
* Contraindication to tocolysis for clinical reasons (e.g. severe pre-eclampsia, chorioamnionitis, placental anomaly, letal fetal anomaly, important intrauterine growth restriction) or current labour
* Contraindication to nifedipine
* Severe renal or hepatic impairment
* Fever > 37.5°C
* Incapacity of communication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Nifedipine blood concentration | Blood collection during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (together with routine blood sampling)
  In total, 3 blood samples are collected after nifedipine administration during hospitalization at the same moment as routine blood sampling. Therefore collection hours are not specified.
Genotyping | Blood collection during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (together with nifedipine blood sampling)
  Pharmacogenetic analysis of genes involved in drug distribution, metabolism and action (e.g. CYP 3A5, POR, CACNA1C) are performed on blood cells of one nifedipine blood sample taken during hospitalization.
Phenotyping | Blood collection during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (together with routine blood sampling)
  Phenotyping of CYP 3A activity is performed during hospitalization by midazolam administration as a probe. Blood is taken at the same moment as routine blood sampling. Therefore collection hour is not specified.

SECONDARY OUTCOMES:
Nifedipine side effects (feeling) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (at 1-3 h after nifedipine administration)
  Nifedipine side effects are collected by questioning patients during hospitalization approximately at 1-3 h after nifedipine administration to assess security of tocolysis (e.g. headache, erythema, nausea).
Maternal heart rate (measurement) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (at 1-3 h after nifedipine administration)
  Maternal heart rate is measured by blood pressure meter during hospitalization approximately at 1-3 h after nifedipine administration to assess security of tocolysis.
Maternal blood pressure (measurement) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (at 1-3 h after nifedipine administration)
  Maternal blood pressure is measured by blood pressure meter during hospitalization approximately at 1-3 h after nifedipine administration to assess security of tocolysis.
Fetal heart rate (measurement) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (during 30-60 min after nifedipine administration)
  Fetal heart rate is measured by cardiotocography during hospitalization approximately during 30-60 min after nifedipine administration to assess security of tocolysis.
Uterine contraction (measurement) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (during 30-60 min after nifedipine administration)
  Uterine contraction is measured by cardiotocography during hospitalization approximately during 30-60 min after nifedipine administration to assess efficacy of tocolysis.
Uterine contraction (feeling) | Evaluation during hospital stay for threatened preterm labour between 20-34 weeks of gestational age (during 2 h after nifedipine administration)
  Frequency and intensity of uterine contraction are collected by questioning patients during hospitalization approximately during 2 h after nifedipine administration to assess efficacy of tocolysis.
Birth date | Data collection after hospital stay for threatened preterm labour between 20-34 weeks of gestational age (potentially at 20-41 weeks of gestational age)
  Time between hospitalization for acute threatened preterm labour and effective birth date is calculated to assess efficacy of tocolysis. This time can be extremely short (inefficacy of tocolysis and delivery in next few hours/days) or correspond to full term.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Panchaud, PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland